CLINICAL TRIAL: NCT04925648
Title: PICAASO / CA180-722: Psma Intensity Can be Altered by Androgen and Phospho-SrC Obstruction
Brief Title: Psma Intensity Can be Altered by Androgen and Phospho-SrC Obstruction
Acronym: PICASSO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St Vincent's Hospital, Sydney (Other)
Responsible Party: Principal Investigator, Anthony Joshua, FRACP, Head of Medical Oncology, The Kinghorn Cancer Centre, St Vincent's Hospital, Sydney
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PICASSO
Record Dates: First submitted 2021-03-23; First posted 2021-06-14 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dasatinib; darolutamide

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomised pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Active Comparator): Dasatinib 100mg once daily orally for 14 Days
  Interventions: Drug: Dasatinib
- Cohort B (Active Comparator): Dasatinib 100mg once daily and Darolumatide 600 mg twice daily orally for 14 Days
  Interventions: Drug: Dasatinib; Drug: Darolutamide

INTERVENTIONS:
Drug: Dasatinib — Dasatinib 100mg once daily orally for 14 Days
Drug: Darolutamide — Darolumatide 600 mg twice daily orally for 14 Days
  Arms: Cohort B

SUMMARY:
The study's purpose is to understand the appearance of your prostate-specific membrane antigen (PSMA) PET scan after you take 14 days of treatment with a drug called dasatinib alone or in combination with anti-testosterone drug call darolutamide.

Who is it for? You may be eligible to join this study if you have metastatic prostate cancer and had a recent PSMA scan showing low PSMA uptake

Study Details:

Participants will receive dasatinib 100 mg daily or dasatinib 100 mg daily and darolutamide 600 mg twice daily for 14 days. They will undergo another PSMA PET scan after 14 days. Participants will be followed up on day 7 of treatment and 30 days after treatment.

It is hoped that this research will provide insight into the mechanism of PSMA expression in advanced prostate cancer.

DETAILED DESCRIPTION:
Our group has previously established a strong interaction between the androgen receptor and PSMA receptor in both castrate sensitive and castrate resistant prostate cancers that impacts on the density of PSMA expression. Recent lab studies have also revealed that phospho-SRC inhibition with drugs such as dasatinib can also modulate PSMA expression, in particular in combination with androgen signalling inhibition. If so, this can influence both the timing and use of PSMA PET scans, PSMA based radionuclide therapies and PSMA immunotherapies. In this study we plan to validate and quantify the change in PSMA PET scan SUV when patients undergo a 14 days treatment with dasatinib alone or in combination with an androgen signalling inhibitor (darolutamide).

ELIGIBILITY:
Inclusion Criteria:

1. Male, aged 18 years or older
2. Pathologically confirmed adenocarcinoma of prostate or a clinical presentation consistent with prostate cancer
3. Metastatic castrate resistant prostate cancer previously confirmed on 68Ga-PSMA-11 and 18F-FDG imaging to be inadequate for future PSMA-directed theranostic treatment by a nuclear medicine physician based on FDG-discordance (FDG-positive, PSMA-negative sites of disease) OR low PSMA SUV values within 2 weeks of starting study drug
4. Adequate hematologic and organ function within 14 days before the first study treatment
5. Castrate levels of testosterone < 1.7 ng/ml
6. Provision of written informed consent.

Exclusion Criteria:

1. Patients who cannot lie still for at least 30 minutes or comply with imaging.
2. Previous dasatinib for prostate cancer or other condition, eg CLL
3. Allergy to dasatinib or darolutamide
4. Use of drugs that interact with interact pharmacologically with dasatinib within 1 week of study entry eg Use of CYP3A4 inducers (e.g. dexamethasone, phenytoin, carbamazepine, rifampicin, phenobarbital or St John's Wort) and use of CYP3A4 substrates with narrow therapeutic index (e.g. astemizole, terfenadine, cisapride, pimozide, quinidine, bepridil or ergot analogues.
5. Use Concomitant use of H2 antagonists or proton pump inhibitors.
6. Current or previous (within the last 6 months) pleural effusion
7. Use of paracetamol during the study period
8. Subjects may not have any of the following: Clinical evidence of uncontrolled heart failure, myocardial infarction, or angina within the previous 6 months; prolonged QT interval Fridericia's (QTcF) > 450msec; history of unstable ventricular arrhythmias (ventricular tachycardia, ventricular fibrillation, or torsades de pointes); concomitant use of drugs known to cause torsades de pointes [quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, dofetilide, erythromycins, clarithromycin, chlorpromazine, haloperidol, mesoridazine,thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl,pentamidine, sparfloxacin, lidoflazine] (these agents must have been discontinued at least 7 days prior to starting dasatinib)
9. Subjects may not be enrolled with any of the following: History of a significant bleeding disorder unrelated to cancer, including diagnosed congenital bleeding disorders (e.g., von Willebrand's disease), and diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies); GI bleeding from any cause within 3 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
To quantify the increase in tumour (standard uptake value) SUV measurements comparing baseline to 2-week PSMA PET scans in men being treated with dasatinib alone or in combination with darolutamide | 14 days
  Primary outcome

SECONDARY OUTCOMES:
To determine the number of participants with treatment-related adverse events as assessed by CTCAE v4.0 after a 14-day course of dasatinib alone or in combination with darolutamide in men with castrate resistant prostate cancer | 14 days
  Secondary outcome

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Kinghorn Cancer Centre, St. Vincent's Hospital, Sydney, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
No Plan to share participant data with individuals outside this trial